CLINICAL TRIAL: NCT00216151
Title: A Randomized Phase II Study of Bisphosphonate: Zoledronic Acid (Zometa) in the Management of Asymptomatic/Early Stage Multiple Myeloma: Hoosier Oncology Group MM02-35
Brief Title: Zoledronic Acid in the Management of Patients With Asymptomatic/Early Stage Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to low patient enrollment.
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Walther Cancer Institute (Other)
Responsible Party: Attaya Suvannasankha, M.D., Hoosier Oncology Group
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HOG MM02-35
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Bisphosphonates
MeSH Terms: conditions — Multiple Myeloma | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Patients will be randomly assigned by study number to receive 4mg of zoledronic acid every three months.
  Interventions: Drug: Zoledronic Acid
- B (No Intervention): Patients will be randomly assigned by study number to observation only.

INTERVENTIONS:
Drug: Zoledronic Acid — Zoledronic Acid 4mg, every three months
  Arms: A

SUMMARY:
Evidence for the beneficial effects of bisphosphonates on bone resorption in multiple myeloma has been reported extensively, showing reductions in skeletal events and improvement of several biochemical variables in bone resorption. Zoledronic acid (Zometa®, CGP42446) is the most potent clinically available bisphosphonates, with the largest therapeutic ratio between the desired inhibition of calcium resorption and the unwanted inhibition of mineralization in vitro of all the bisphosphonates.

This trial will investigate the efficacy of zoledronic acid in preventing skeletal events in patients with asymptomatic/early stage Multiple Myeloma

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

* Patients will be randomly assigned by study number to receive 4mg of zoledronic acid every three months or to be observed.

Performance status: ECOG performance status 0-3 (KPS 30 - 100)

Life expectancy: 12 months

Hematopoietic:

* Hb >10 g/dl within 14 days prior to registration

Hepatic:

* Not specified

Renal:

* Serum creatinine < 2 mg/dl within 14 days prior to registration

Cardiovascular:

* Not specified

Pulmonary:

* Not specified

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asymptomatic multiple myeloma as defined by the criteria below:
* Presence of bone marrow clonal plasma cells (more than 10%)
* Presence of an M-protein in serum and/or urine (no concentration specified)
* Serum calcium < 12 mg/dl within 14 days prior to registration. Less than 3 lytic lesions, no pathologic fractures and no osteopenia noted on skeletal survey
* No symptoms of hyperviscosity, amyloidosis or recurrent infection
* Bone mineral density with a T score higher than -2.0 standard deviation (not have osteoporosis) within 28 days prior to registration
* Negative pregnancy test

Exclusion Criteria:

* No previous treatment with bisphosphonates
* No disorders of the parathyroid or thyroid glands
* No current breastfeeding
* No prior malignancy is allowed except for adequately treated in situ cervical cancer, Gleason < grade 7 prostate cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2005-06; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
· To examine the effect of intravenous zoledronic acid at the dose of 4 mg given every three months compared with observation, on percent change in bone mineral density of the spine at one year in patients with asymptomatic, smoldering and stage I MM. | 18 months

SECONDARY OUTCOMES:
· To examine the effect of intravenous zoledronic acid at the above schedule on percent change in bone mineral density of the total hip and femur. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Attaya Suvannasankha, M.D., Study Chair — Hoosier Oncology Group, LLC
Locations (8):
- United States (8):
  - Elkhart Clinic, Elkhart, Indiana
  - Oncology Hematology Associates of SW Indiana, Evansville, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Quality Cancer Center (MCGOP), Indianapolis, Indiana
  - Arnett Cancer Care, Lafayette, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Providence Medical Group, Terre Haute, Indiana
  - AP&S Clinic, Terre Haute, Indiana

REFERENCES:
- See also: Hoosier Oncology Group Home Page — http://hoosieroncologygroup.org/